CLINICAL TRIAL: NCT01412515
Title: A Phase II Study With Tumor Molecular Pharmacodynamic (MPD) Evaluation of Oral mTOR-inhibitor Everolimus (RAD001) 10 mg Daily in Patients Suffering From Classic or Endemic Kaposi's Sarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: results from interim analysis conducted to study interruption
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C06-46
Record Dates: First submitted 2011-08-08; First posted 2011-08-09 (Estimated); Last update posted 2012-01-02 (Estimated); Status verified 2011-08

CONDITIONS: Kaposi Sarcoma
Keywords: mTOR inhibitors
MeSH Terms: conditions — Sarcoma, Kaposi | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus (Experimental): everolimus 10 mg per day
  Interventions: Drug: everolimus

INTERVENTIONS:
Drug: everolimus — everolimus per os 10mg per day

SUMMARY:
Classic Kaposi's sarcoma (CKS) is an angioproliferation associated with human herpes virus 8 (HHV8), which sometimes requires systemic treatment. Rapamycin and everolimus are mTOR inhibitors. The PI3K-AKT-mTOR pathway is activated in CKS.The aim of this study is to evaluate the rate of clinical response and tolerance to everolimus 10mg/d in CKS. Patients suffering from CKS will be enrolled in a multicenter two-stage phase II trial. At inclusion, all patients will have at least 10 lesions or more than one limb or 3% of body surface affected, in the absence of symptomatic visceral CKS. The primary endpoint is objective response to everolimus after 6 months therapy (complete or partial response per ACTG criteria). The trial is planned using Simon's minimax two-stage design to demonstrate a response rate of 50% as compared to 20% with type I error rate 2.5% and power of 90%. Accordingly, 11 patients will to be enrolled in the first stage and provided at least 3 patients responded, 15 patients will be accrued in a second stage.

DETAILED DESCRIPTION:
The primary endpoint is objective response to everolimus after 6 months therapy (complete or partial response per ACTG criteria).

Secondary endpoints are response according to physician global assessment, lesions size , lesions infiltration, lymphedema, tolerance, pharmacodynamic (pathologic, angiogenic and lymphangiogenic biomarkers, HHV8 viral load sequential evaluation in the lesions, pharmacokinetic evaluation.

ELIGIBILITY:
Inclusion Criteria:

Histologic confirmed classic or endemic KS (non transplant non HIV patients) > 18 Years old at least 10 lesions or more than one limb or 3% of body surface affected, in the absence of symptomatic visceral KS Presence of at least 4 targets lesions > 5mm At least 4 weeks wash out from any KS specific therapy ECOG < 2

Exclusion Criteria:

immunosupressive regimen patients HIV positive creatinine clearance <40ml/mn,AST ALT>3N, neutropénia<1500, thrombopenia<150000, anemia<8g/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
objective response to everolimus after 6 months therapy | duration of study 30 months
  objective response to everolimus after 6 months therapy (complete or partial response per ACTG criteria).

SECONDARY OUTCOMES:
response according to physician global assessment, lesions size , lesions infiltration | 30 months
  response according to physician global assessment, lesions size , lesions infiltration

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Lebbé, MD, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Hospital Saint Louis, Paris, France